CLINICAL TRIAL: NCT00950456
Title: A Prospective Non-Interventional Observational Study to Assess the Safety of Two Vaccinations of a Vero Cell-Derived, Whole Virus H1N1 Pandemic Influenza Vaccine in Subjects Exposed to the Vaccine Through Policies by Governments or Health Authorities
Brief Title: Observational Study to Assess Safety of H1N1 Pandemic Influenza Vaccine
Status: Completed | Type: Observational
Sponsor: Alachua Government Services, Inc. (Industry)
Responsible Party: David Perry, MD; Sponsor´s signatory, Baxter Innovations GmbH
Other Study IDs: 820901
Record Dates: First submitted 2009-07-30; First posted 2009-07-31 (Estimated); Last update posted 2015-10-09 (Estimated); Status verified 2011-05

CONDITIONS: Influenza; Pandemic Influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- H1N1 Pandemic Influenza Vaccine: Subjects will be enrolled and vaccinated according to national policy and standard practice.
  Interventions: Biological: H1N1 Pandemic Influenza Vaccine (whole virion, Vero Cell-derived, inactivated)

INTERVENTIONS:
Biological: H1N1 Pandemic Influenza Vaccine (whole virion, Vero Cell-derived, inactivated) — It is anticipated that subjects will receive two intramuscular injections approximately 3 weeks apart. The vaccine will be provided in two doses, one for adults, the other for children.
  Other Names: CELVAPAN

SUMMARY:
The purpose of this observational study, which will be initiated as soon as the licensed H1N1 Pandemic Influenza Vaccine is used in a mass vaccination campaign, is to estimate the incidence of any medically-attended adverse events in all vaccinated subjects.

ELIGIBILITY:
Inclusion Criteria:

Male and female subjects, per indication on license or per official vaccine recommendations, will be eligible for participation in this study if:

* They will be administered CELVAPAN (= Baxter´s H1N1 pandemic influenza vaccine)
* They are 2 months of age or older at the time of first vaccine administration
* Their medical history is available
* The investigator believes they will comply with the foreseen vaccination schedule and will reliably observe signs or symptoms of adverse events during the observational period
* They and/or their parent(s)/legal guardian(s) provide written informed consent, and assent where appropriate, prior to study entry according to national law

Exclusion Criteria:

Male and female subjects will be excluded from participation in this study if:

* They have already been administered another H1N1 pandemic vaccine
* They have any contraindication to vaccination (as per the Summary of Product Characteristics and/or relevant national immunization guidelines)

Min Age: 2 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The enrollment of subjects in this study will follow national vaccination policy decisions in the UK.
Sampling Method: Non-Probability Sample
Enrollment: 3216 (Actual)
Dates: Start 2009-11; Primary Completion 2010-12 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Baxter BioScience Medical Director, Study Director — Baxter Healthcare Corporation
Locations (17):
- Austria (17):
  - General Practice, Bludenz
  - General Practice, Fulpmes
  - General Practice, Hall in Tirol
  - General Practice, Innsbruck
  - Practice for Travel Medicine, Innsbruck
  - City Council (Magistrat) Klagenfurt (Health & Food Department), Klagenfurt
  - General Practice, Kufstein
  - General Practice, Mariapfarr
  - General Practice, Oberperfuss
  - General Practice, Salzburg
  - General Practice, Telfs
  - Medical University of Vienna, Department of Internal Medicine I, Division of Infectious Diseases and Tropical Medicine, Vienna
  - Medical University of Vienna, Department of Specific Prophylaxis and Tropical Medicine, Vienna
  - Hanusch Hospital, Vienna
  - Wiener Gebietskrankenkasse (Health insurance center Vienna), Vienna
  - General Practice, Voitsberg
  - General Practice, Wels